CLINICAL TRIAL: NCT05162976
Title: A Phase 1 Study of CC-486 Plus Nivolumab in Patients With Hodgkin Lymphoma Refractory to PD-1 Therapy
Brief Title: CC-486 and Nivolumab for the Treatment of Hodgkin Lymphoma Refractory to PD-1 Therapy or Relapsed
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21319; P30CA033572 (NIH); NCI-2021-13436 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 21319 (Other: City of Hope Medical Center)
Record Dates: First submitted 2021-12-16; First posted 2021-12-20 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Recurrent Classic Hodgkin Lymphoma; Refractory Classic Hodgkin Lymphoma
MeSH Terms: interventions — Nivolumab; Azacitidine; cc-486

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (CC-486, nivolumab) (Experimental): Patients receive azacitidine PO QD on days 1-7 and nivolumab IV over 30 minutes on day 8. Treatment repeats every 28 days for up to 24 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Nivolumab; Drug: Oral Azacitidine

INTERVENTIONS:
Biological: Nivolumab — Given IV
  Other Names: BMS-936558; CMAB819; MDX-1106; NIVO; Nivolumab Biosimilar CMAB819; ONO-4538; Opdivo
Drug: Oral Azacitidine — Given PO
  Other Names: CC-486

SUMMARY:
This phase I trial tests the safety and best dose of CC-486 (an oral form of azacitidine) when given together with nivolumab in treating patients with Hodgkin lymphoma that does not respond (refractory) to PD1-based immunotherapy or has come back (relapsed). CC-486 is in a class of medications called demethylation agents. It works by helping the bone marrow to produce normal blood cells and by killing abnormal cells. Immunotherapy with monoclonal antibodies, such as nivolumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Giving CC-486 in combination with nivolumab may render nivolumab more effective.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Evaluate the safety and tolerability of a regimen combining oral azacitidine (CC-486) and nivolumab in patients with Hodgkin lymphoma (HL) refractory to PD1/PD-L1 therapy.

II. Estimate the overall response rate (ORR) in patients treated with CC-486 plus nivolumab.

SECONDARY OBJECTIVE:

I. Estimate the complete response (CR) rate, duration of response (DOR), progression-free survival (PFS) and overall survival (OS) in patients treated with CC-486 plus nivolumab.

EXPLORATORY OBJECTIVES:

I. Examine the association between clinical outcomes with nivolumab + CC-486 and circulating tumor-derived deoxyribonucleic acid (ctDNA) characteristics (mutation profile, kinetics of clearance).

II. Examine changes in peripheral blood immune subsets, clonality, and T-cell receptor (TCR) repertoire during treatment with nivolumab and CC-486.

III. Examine the pre-treatment cellular spatial relationships in the tumor microenvironment by geographical mapping and assess association with response.

IV. Explore the association between baseline total metabolic tumor volume, complete response, and PFS after CC-486 plus nivolumab therapy.

V. Explore the association between change in total metabolic tumor volume between baseline and 16 weeks, complete response, and PFS after CC-486 plus nivolumab therapy.

VI. Explore the association between outcomes (overall response, complete response, PFS) and other baseline quantitative positron emission tomography (PET) (qPET) parameters including total lesion glycolysis and standardized uptake value maximum (SUVmax).

OUTLINE: This is a dose-expansion study of azacitidine.

Patients receive azacitidine orally (PO) once daily (QD) on days 1-7 and nivolumab intravenously (IV) over 30 minutes on day 8. Treatment repeats every 28 days for up to 24 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days, every 12 weeks for 1 years, and then every 24 weeks for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Documented informed consent of the participant and/or legally authorized representative

  * Assent, when appropriate, will be obtained per institutional guidelines
* Be willing to provide tissue from a fresh core or excisional biopsy (performed as standard of care) of a tumor lesion prior to starting study therapy or from archival tissue of a biopsy that was performed after the most recent systemic therapy

  * Exception may be granted by the principal investigator (PI) if a biopsy is not feasible and/or safe
* Age: >= 18 years
* Eastern Cooperative Oncology Group (ECOG) =< 2
* Histologically confirmed diagnosis of classical Hodgkin lymphoma (excluding nodular lymphocyte predominant Hodgkin lymphoma) according to the World Health Organization (WHO) classification, with hematopathology review at the participating institution
* Refractory to PD-1/PD-L1 directed immunotherapy, defined as patients who had prior exposure to PD-1/PD-L1 immunotherapy and either:

  * Achieved a best response of PD, or
  * Achieved a best response of CR/PR but developed PD while on active PD-1/PD-L1 treatment or within 12 weeks of last dose of PD-1/PD-L1 treatment
* Relapse must have been confirmed histologically (with hematopathology review at the participating institution)

  * Exceptions may be granted with study PI approval
* Patient must have received at least one prior systemic therapy and must not currently be candidate for stem cell transplantation
* Measurable disease by computed tomography (CT) or positron emission tomography (PET)/CT scan with one or more sites of disease >= 1.5 cm in longest dimension
* Fully recovered from the acute toxic effects (except alopecia) to =< Grade 1 to prior anti-cancer therapy
* Absolute neutrophil count (ANC) >= 1,000/mm^3

  * NOTE: Growth factor is not permitted within 7 days of ANC assessment unless cytopenia is secondary to disease involvement
* Platelets >= 75,000/mm^3

  * NOTE: Platelet transfusions are not permitted within 7 days of platelet assessment unless cytopenia is secondary to disease involvement
* Hemoglobin >= 8 g/dL
* Total bilirubin =< 1.5 x upper limit of normal (ULN) or =< 3 x ULN if patient has Gilbert's disease OR direct bilirubin =< ULN for subjects with total bilirubin levels > 1.5 x ULN
* Aspartate aminotransferase (AST) =< 2.5 x ULN OR =< 5 x ULN for subjects with liver involvement by lymphoma as the etiology of transaminase elevation
* Alanine aminotransferase (ALT) =< 2.5 x ULN OR =< 5 x ULN for subjects with liver involvement by lymphoma as the etiology of transaminase elevation
* Creatinine clearance of >= 40 mL/min per 24 hour urine test or the Cockcroft-Gault formula
* If not receiving anticoagulants: International normalized ratio (INR) OR prothrombin (PT) =< 1.5 x ULN

  * If on anticoagulant therapy: PT must be within therapeutic range of intended use of anticoagulants
* If not receiving anticoagulants: Activated partial thromboplastin time (aPTT) =< 1.5 x ULN

  * If on anticoagulant therapy: aPTT must be within therapeutic range of intended use of anticoagulants
* Women of childbearing potential (WOCBP): negative urine or serum pregnancy test

  * If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Agreement by females and males of childbearing potential* to use an effective method of birth control or abstain from heterosexual activity for the course of the study through at least 5 months after the last dose of nivolumab and 6 months after the last dose of CC-486 for females, and 3 months after the last dose of CC-486 for males with female partners of reproductive potential

  * Childbearing potential defined as not being surgically sterilized (men and women) or have not been free from menses for > 1 year (women only)

Exclusion Criteria:

* Prior allogeneic stem cell transplant within 6 months prior to day 1 of protocol therapy
* If prior allogeneic transplant, then no active graft-versus-host disease (GVHD), no systemic immunosuppression for at least 3 months prior to study enrollment, and no history of grade 3-4 acute GVHD
* Autologous stem cell transplant within 3 months prior to day 1 of protocol therapy
* Prior solid organ transplant
* Systemic steroid therapy for lymphoma symptom control must be tapered down to =< 10 mg/day prednisone or equivalent
* Live vaccine within 30 days prior to day 1 of protocol therapy
* Concomitant investigational therapy
* History of prior >= grade 3 hypersensitivity to nivolumab, or history of allergic reactions attributed to compounds of similar chemical or biologic composition to study agents or to any of the excipients, including mannitol
* Known active central nervous system (CNS) involvement by lymphoma
* History of active pneumonitis or interstitial lung disease requiring supplemental oxygen or corticosteroid treatment
* History of inflammatory bowel disease (e.g., Crohn's disease, ulcerative colitis), celiac disease (i.e., sprue), prior gastrectomy or upper bowel removal, or any other gastrointestinal disorder or defect that would interfere with the absorption, distribution, metabolism or excretion of the study drug and/or predispose the subject to an increased risk of gastrointestinal toxicity
* History of another primary malignancy that has not been in remission for at least 2 years, with the following exceptions:

  * Adequately treated non-melanoma skin cancer or lentigo maligna (melanoma in situ) without evidence of disease
  * Adequately treated in situ carcinomas (e.g. cervical, esophageal) without evidence of disease
  * Asymptomatic prostate cancer managed with a watch-and-wait strategy
  * If the malignancy is expected to not require any treatment for at least 2 years (this exception should be discussed with the study PI)
* History of progressive multifocal leukoencephalopathy (PML)
* Prior diagnosis of inherited or acquired immunodeficiency
* Active, known or suspected autoimmune disease. The following are exceptions:

  * Vitiligo
  * Psoriasis not requiring systemic treatment
  * Hemolytic anemia associated with the lymphoma
  * Type I diabetes mellitus, if adequately controlled with therapy
  * Thyroid disease, if adequately controlled with therapy

    * Any autoimmune disease should have not been treated with systemic disease-modifying antirheumatic drugs for the last 2 years. All patients with a history of autoimmune disease except for the above should be discussed with the study PI
* Uncontrolled systemic fungal, bacterial or viral infection (defined as ongoing signs/symptoms related the infection without improvement despite appropriate antibiotics, antiviral therapy and/or other treatment)
* Clinically significant uncontrolled illness
* History of a cerebral vascular event (stroke or transient ischemic attack), unstable angina, myocardial infarction, or cardiac symptoms consistent with New York Heart Association Class III-IV within 6 months prior to day 1 of protocol therapy
* Known active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection. Patients with past HBV infection (defined as negative hepatitis B surface antigen [HBsAg] and positive hepatitis B core antibody [HBcAb]) are eligible if HBV deoxyribonucleic acid (DNA) is undetectable. Patients who are positive for HCV antibody are eligible if polymerase chain reaction (PCR) is negative for HCV ribonucleic acid (RNA). Testing to be done only in patients suspected of having infections or exposures
* Known active human immunodeficiency virus (HIV) infection. Subjects who have an undetectable or unquantifiable HIV viral load with CD4 > 200 and are on highly active antiretroviral therapy (HAART) medication are allowed. Testing to be done only in patients suspected of having infections or exposures
* Females only: Pregnant or breastfeeding
* Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2022-01-03 (Actual); Primary Completion 2026-05-12 (Estimated); Study Completion 2026-05-12 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity | Up to 28 days (1 cycle)
  Toxicities will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events ([CTCAE], version 5.0).
Overall response rate (ORR) | Up to 2 years
  Defined as the proportion of patients that have a documented complete response (CR) or particle response (PR) at any time during study treatment. Will be estimated by the proportion of response-evaluable patients achieving CR or PR along with the 95% exact binomial confidence interval.

SECONDARY OUTCOMES:
Complete response (CR) rate | Up to 2 years
  Defined as the proportion of patients that have a documented CR at any time during study treatment.
Duration of response (DOR) | Up to 2 years
  Will be estimated using the product-limit method of Kaplan and Meier along with the Greenwood estimator of standard error; 95% confidence interval will be constructed based on log-log transformation. Median DOR will be estimated when available.
Overall survival (OS) | Time from initiation of study therapy to death from any cause, assessed up to 2 years
  Will be estimated using the product-limit method of Kaplan and Meier along with the Greenwood estimator of standard error; 95% confidence interval will be constructed based on log-log transformation. Median OS will be estimated when available.
Progression-free survival (PFS) | Time from initiation of study therapy to the first observation of disease relapse/progression or death from any cause, whichever occurs first, assessed up to 2 years
  Will be estimated using the product-limit method of Kaplan and Meier along with the Greenwood estimator of standard error; 95% confidence interval will be constructed based on log-log transformation. Median PFS will be estimated when available.
Incidence of adverse events | Up to 30 days after last dose
  Toxicity and adverse events will be recorded using the National Cancer Institute (NCI) CTCAE 5.0 scale.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Mei, MD, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States